CLINICAL TRIAL: NCT00818688
Title: Superficial Thrombophlebitis and Venous Thromboembolism: A Large Prospective Epidemiological Study
Brief Title: POST (Prospective Observational Superfial Thrombophlebitis)
Acronym: POST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Pr DECOUSUS Hervé, CHU de SAINT-ETIENNE
Other Study IDs: 0401080
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Thrombophlebitis
Keywords: Superficial thrombophlebitis (ST); Deep-vein thrombosis; Symptomatic pulmonary embolism; Symptomatic Superficial Thrombophlebitis of the lower limbs
MeSH Terms: conditions — Thrombophlebitis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients eligible for enrolment were all consecutive patients aged 18 years or over, with a symptomatic ST of the lower limbs at least 5 cm long on compression ultrasonography. Patients who had undergone surgery under general or loco-regional anaesthesia in the previous 10 days, those in whom ST had occurred after sclerotherapy within the previous 30 days and those whose follow-up was not considered to be feasible were ineligible.
  Interventions: Procedure: compression ultrasonography at 3 months
- 2: Patients eligible for enrolment were all consecutive patients aged 18 years or over, with a symptomatic ST of the lower limbs at least 5 cm long on compression ultrasonography. Patients who had undergone surgery under general or loco-regional anaesthesia in the previous 10 days, those in whom ST had occurred after sclerotherapy within the previous 30 days and those whose follow-up was not considered to be feasible were ineligible.

INTERVENTIONS:
Procedure: compression ultrasonography at 3 months — A three-month follow-up prospective study was performed in the subgroup of patients with symptomatic ST but without deep-vein thrombosis on compression ultrasonography or documented symptomatic pulmonary embolism at inclusion, a group defined as patients with 'isolated ST'.
  Groups: 1

SUMMARY:
We performed a national cross-sectional and prospective large epidemiological cohort study in patients with ST. Office- and hospital-based vascular medicine French practitioners enrolled all consecutive patients with a symptomatic ST of the lower limbs at least 5 cm long documented by compression ultrasonography. Follow-up was three months. All events were adjudicated by a central committee.

DETAILED DESCRIPTION:
Between March 2005 and October 2006, 844 patients (median age [range]: 65 [18-98] years; 547 women) were included. At inclusion, confirmed deep-vein thrombosis and/or symptomatic pulmonary embolism was associated with ST in 24.9% (n=210) of patients. Among the 600 patients with isolated ST (i.e. without deep-vein thrombosis or pulmonary embolism at inclusion), 10.4% (n=56) developed venous thromboembolic complications at three months, including the following symptomatic events: pulmonary embolism (0.4%, n=2), deep-vein thrombosis (2.8%, n=15), extension of ST (3.1%, n=17) and recurrence of ST (1.9%, n=10). These complications occurred despite the use of various anticoagulant strategies in 90.5% (n=540) of patients; four independent risk factors increased the risk of these complications: male sex, cardiac or respiratory insufficiency, history of deep-vein thrombosis or pulmonary embolism and no history of varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients aged 18 years or over, with a symptomatic ST of the lower limbs at least 5 cm long on compression ultrasonography.

Exclusion Criteria:

* patients who had undergone surgery under general or loco-regional anaesthesia in the previous 10 days, those in whom ST had occurred after sclerotherapy within the previous 30 days and those whose follow-up was not considered to be feasible were ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ST of the lower limbs.
Sampling Method: Non-Probability Sample
Enrollment: 844 (Actual)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence of confirmed venous thromboembolism at three months. | 3 months

SECONDARY OUTCOMES:
Overall mortality at three months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DECOUSUS, Pr, Principal Investigator — CHU de SAINT-ETIENNE
Locations (5):
- France (5):
  - LEANDRI, Annonay
  - CHANUT, Aubenas
  - GILLET, Bourgoin Jailleu
  - Barrelier, Caen
  - Guenneguez, Dieppe

REFERENCES:
- [Derived] Galanaud JP, Bosson JL, Genty C, Presles E, Cucherat M, Sevestre MA, Quere I, Decousus H, Leizorovicz A. Superficial vein thrombosis and recurrent venous thromboembolism: a pooled analysis of two observational studies. J Thromb Haemost. 2012 Jun;10(6):1004-11. doi: 10.1111/j.1538-7836.2012.04704.x. PMID 22429908
- [Derived] Decousus H, Quere I, Presles E, Becker F, Barrellier MT, Chanut M, Gillet JL, Guenneguez H, Leandri C, Mismetti P, Pichot O, Leizorovicz A; POST (Prospective Observational Superficial Thrombophlebitis) Study Group. Superficial venous thrombosis and venous thromboembolism: a large, prospective epidemiologic study. Ann Intern Med. 2010 Feb 16;152(4):218-24. doi: 10.7326/0003-4819-152-4-201002160-00006. PMID 20157136